CLINICAL TRIAL: NCT01553292
Title: Feasibility of Using Early CPAP (Continuous Positive Airway Pressure) And Large Volume Minimal Invasive Surfactant Therapy (ECALMIST) in Preterm Infants With Respiratory Distress Syndrome (RDS)
Brief Title: Early CPAP And Large Volume Minimally Invasive Surfactant (ECALMIST) in Preterm Infants With RDS
Acronym: ECALMIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Yahya Al Ethawi, Principal Investigator MD, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2012:016
Record Dates: First submitted 2012-03-06; First posted 2012-03-14 (Estimated); Results first posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-06

CONDITIONS: Respiratory Distress Syndrome
Keywords: Respiratory distress syndrome; Preterm infants; Vascular catheter; Surfactant; CPAP; ECALMIST
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ECALMIST (Experimental): Large volume 5ml/kg surfactant administered by vascular catheter while maintaining CPAP or ECALMIST; Early CPAP (continuous positive airway pressure) And Large volume Minimal Invasive Surfactant Therapy
  Interventions: Device: ECALMIST

INTERVENTIONS:
Device: ECALMIST — Labelled catheter at level of the lips (6 cm plus weight) will inserted through the vocal cords under direct vision using a standard laryngoscope without premedication while maintaining CPAP. 5 ml/kg surfactant syringe will be connected to the catheter hub and 0.25-0.5 ml was administered; then the syringe will be disconnected from the catheter to observe the surfactant moving up and down or coming back as indication of accurate intubation of the trachea. The surfactant the slowly administer by boluses of 0.25-0.5 ml over 20-30 seconds with 10 seconds apart. At the end of the procedure, the operator flushed the catheter with 0.5 ml of air before removing the catheter while maintaining CPAP
  Other Names: Surfactant administration by catheter
Device: ECALMIST — Vascular catheter of 1.6 French size of 133 mm length 16 gauge used to deliver the BLES; a large volume surfactant while maintain CPAP
  Other Names: Surfactant administration by catheter

SUMMARY:
Modification of Minimally Invasive Surfactant Therapy (MIST) to a new technique called ECALMIST (Early CPAP And Large volume Minimal Invasive Surfactant). This modification is needed to adapt the use of large volume surfactant of 4-5 ml/kg.

The ECALMIST will be used to deliver the large volume Surfactant that been used in Canada called BLES (about 5 ml for each 100 mg) to the preterm infants bellow 35 weeks gestation suffer from respiratory distress syndrome (RDS) in 1st 24 hours of life while maintained on CPAP.

DETAILED DESCRIPTION:
The 5 ml/Kg surfactant is warm to room temperature. Using standard laryngoscope without premedication while the infant is maintained on continuous positive airway pressure (CPAP. The the laryngoscope should be removed after stabilizing the vascular catheter between 2 fingers at the level of lips (weight +6 cm). The surfactant will be administer by boluses of 0.25 -0.5 ml at a time over 20-30 seconds and 10 seconds apart while maintain the vital signs.

The procedure should be stopped if the vital signs deteriorate, CPAP pressure and oxygen requirement might need to adjusted to restore baseline vital signs. If the vital signs remained unstable the catheter should be removed and the infant managed according by positive pressure ventilation (PPV) or intubation by endotracheal tube (ETT).

At the end of the procedure the catheter should be flushed with 0.5 ml of air then catheter should be removed.

FiO2 (fraction of inspired oxygen), oxygen saturation and CPAP pressure will be recorded before during and after the procedure.

Complication like bradycardia (Hear rate below 100 beat per minute) or Apnea (pause of respiration for more than 20 second or less than 20 seconds but associated with bradycardia) All other neonatal outcome will be recorded (IVH [Intra-ventricular Hemorrhage], ROP [Retinopathy of prematurity], duration of ventilation, duration of hospital stay, infection, duration of oxygen requirement and others.

ELIGIBILITY:
Inclusion Criteria:

-preterm infants less than 35 weeks gestation in 1st day of life with RDS and spontaneously breathing on CPAP and need surfactant administration.

Exclusion Criteria:

* Infants needs of mechanical ventilation
* Congenital anomaly
* Respiratory distress due to non RDS related causes.
* no parental consent

Ages: 10 Minutes to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yahya Al Ethawi, MD, Principal Investigator — University of Manitoba
Locations (3):
- Canada (3):
  - Children hospital of health Sciences Center, Winnipeg, Manitoba
  - Women's Hospital Health Science Center, Winnipeg, Manitoba
  - St. Boniface Hospital, Winnipeg, Manitoba

REFERENCES:
- See also: If parents, colleagues have any questions, comments or suggestions; you can contact me on Facebook with this link — http://www.facebook.com/yahya.alethawi?sk=notes#!/?sk=nf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was of 2 months duration form July 5th, 2012 to September 5th, 2012 in 3 hospitals (St Boniface NICU, Children hospital's NICU and Women's hospital delivery room at HSC).
Groups:
- Surfactant Through Vascular Catheter: Preterm infants born between 24 to 34 weeks postmenstrual gestation were received surfactant by using technique called ECALMIST (Early CPAP And Large Volume Minimal Invasive Surfactant)during 1st 24 hours of life
Period: Overall Study
Arm/Group | Surfactant Through Vascular Catheter
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Angiocath Surfactant: Preterm infants born at 24 to 34 weeks of postmenstrual gestational age were received surfactant by using technique called ECALMIST (Early CPAP And Large Volume Minimal Invasive Surfactant)
Arm/Group | Angiocath Surfactant
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: Weeks] | 29 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Region of Enrollment [Number; unit: participants]
  Canada | 21

OUTCOME MEASURES:

1. Secondary Outcome: Incidence of Bradycardia During Procedure
Description: Bradycardia is persistent heart rate below 100 beat per minute for more than 20 seconds during the procedure as seen by the monitor or Heart rate below 60 beat per minute for any time if chest compression is needed or if associated with desaturation or apnea.
Time Frame: Range of 10 minutes
Population: The mean of heart beat per minute of all participants during ECALMIST(measured by minutes which is variable according participant tolerance of the ECALMIST procedure)
Measure: Number; unit: Number of participants
Groups:
- Surfactant Administration Through Vascular Catheter: Preterm infants from 24 to 34 weeks were received surfactant by using technique called ECALMIST (Early CPAP And Large Volume Minimal Invasive Surfactant)
Arm/Group | Surfactant Administration Through Vascular Catheter
Number analyzed (Participants) | 21
Number of participants | 3

2. Secondary Outcome: Saturation During the Procedure
Description: Level of oxygen which is measured by oxygen pulse Oximetry. It is express as proportion out of one which is equal to percentage of 100. The number can be anywhere between 0.21 to 1 which is equal to percentage of 21 to 100.
Time Frame: 10 minutes
Population: The mean of oxygen saturation of all participants during ECALMIST(measured by minutes which is variable according participant tolerance of the ECALMIST procedure)
Measure: Mean (Standard Deviation); unit: Proportion of oxygen saturation
Groups:
- Surfactant Administration Through Vascular Catheter: Preterm infants born between 24 to 34 weeks post-menstrual age were received surfactant by using technique called ECALMIST (Early CPAP And Large Volume Minimal Invasive Surfactant)
Arm/Group | Surfactant Administration Through Vascular Catheter
Number analyzed (Participants) | 21
Proportion of oxygen saturation | 0.87 (0.08)

3. Secondary Outcome: Failure to Catheterized the Trachea by the Vascular Catheter
Description: Failure define as inability to pass the vascular catheter to the trachea after 2 trials within 20 seconds time frame for each trial.
Time Frame: 20 seconds
Population: Number of infatns that failed to pass the angiocath to the trachea after 2 trials, 20 seconds each trial.
Measure: Number; unit: Number of participants
Arm/Group | Surfactant Administration Through Vascular Catheter
Number analyzed (Participants) | 21
Number of participants | 1

4. Primary Outcome: Incidence of Early Ventilation Hours
Description: The need for mechanical ventilation due to various reasons like sepsis, Apnea (pause of respiration for more than 20 seconds) or Respiratory dysfunction evidenced by abnormal blood gas or desaturation or increase work of breathing
Time Frame: 72 hours
Population: The number of preterm infants that need intubation by ETT within 72 hours of life(early ventilation). This is includes all infants intubated whether during or after the ECALMIST procedure in the 1st 3 days of life (after delivery)
Measure: Number; unit: Number of participants
Arm/Group | Surfactant Administration Through Vascular Catheter
Number analyzed (Participants) | 21
Number of participants | 4

5. Secondary Outcome: Index Before the Procedure
Description: The index is an arbitrary number calculated by equation that is author defined which is(FiO2 * CPAP/ Sat)*100.
  FiO2: Fraction of inspired oxygen CPAP: continuous positive airway pressure Sat: saturation The equation is similar to the Oxygen index (OI) equation with replacement of Mean airway pressure (MAP) by continuous positive airway pressure (CPAP. It comprehensive view about the 3 parameters (FiO2, CPAP and Sat) during the procedure.
Time Frame: 1 hour
Population: The mean of index of all participants before ECALMIST
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Surfactant Administration Through Vascular Catheter: Preterm infants between 24 to 34 weeks were received surfactant by using technique called ECALMIST (Early CPAP And Large Volume Minimal Invasive Surfactant)
Arm/Group | Surfactant Administration Through Vascular Catheter
Number analyzed (Participants) | 21
Score | 2.61 (0.81)

6. Secondary Outcome: CPAP Pressure After the Procedure
Description: Continuous positive airway pressure (CPAP) is measured in centimeter of water
Time Frame: 4 hours
Population: The mean of CPAP pressure express as centimeter of water of all participants after completion of ECALMIST
Measure: Mean (Standard Deviation); unit: Centimeter of water
Arm/Group | Surfactant Administration Through Vascular Catheter
Number analyzed (Participants) | 21
Centimeter of water | 5.8 (0.471)

7. Secondary Outcome: Oxygen Requirement Before the Procedure
Description: Oxygen requirement or FiO2 (Fraction of inspired oxygen) is expressed as proportion out of one (decimal) or percentage of 100. The number can be any where between 0.21 to 1 which is equal to percentage of 21 to 100.
Time Frame: 1 hour
Population: The mean of oxygen requirement of all the participants before ECALMIST
Measure: Mean (Standard Deviation); unit: Proportion of oxygen requirement
Arm/Group | Surfactant Administration Through Vascular Catheter
Number analyzed (Participants) | 21
Proportion of oxygen requirement | 0.308 (0.068)

8. Secondary Outcome: Oxygen Saturation After the Procedure
Description: Oxygen saturation is measured by pulse oximetry. It is express as proportion out of 1 (decimal) that is equal to percentage of 100. The number can be any where between 0.21 to 1 which is equal to percentage of 21 to 100.
Time Frame: 4 hours
Population: The mean of oxygen saturation after ECALMIST for all the participants
Measure: Mean (Standard Deviation); unit: Proportion of oxygen saturation
Arm/Group | Surfactant Administration Through Vascular Catheter
Number analyzed (Participants) | 21
Proportion of oxygen saturation | 0.94 (0.04)

9. Secondary Outcome: Index After the Procedure
Description: as for outcome 5
Time Frame: 4 hours
Population: The mean of ECALMIST index of all the participants after ECALMIST
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Surfactant Administration Through Vascular Catheter
Number analyzed (Participants) | 21
Score | 1.27 (1.8)

10. Secondary Outcome: CPAP Pressure Before the Proceudre
Description: Continuous positive airway pressure (CPAP) pressure is measured in centimeter of water as recorded from CPAP machine (continuous positive airway pressure)
Time Frame: 1 hour
Population: The mean of CPAP pressure that is measured by centimeter of water of all the participant before ECALMIST
Measure: Mean (Standard Deviation); unit: Centimeter of water
Arm/Group | Surfactant Administration Through Vascular Catheter
Number analyzed (Participants) | 21
Centimeter of water | 7.1 (0.447)

11. Secondary Outcome: Oxygen Saturation Before the Procedure
Description: Oxygen saturation is measured by pulse oximetry and express as proportion out of one which equal to percentage of 100. The number can be any where between 0.21 to 1 which is equal to percentage of 21 to 100.
Time Frame: 1 hour
Population: The mean of saturation of all participants before ECALMIST
Measure: Mean (Standard Deviation); unit: Proportion of oxygen saturation
Arm/Group | Surfactant Administration Through Vascular Catheter
Number analyzed (Participants) | 21
Proportion of oxygen saturation | 0.87 (0.08)

12. Secondary Outcome: Oxygen Requirements After the Procedure
Description: Oxygen requirement is expressed as proportion out of one (decimal) which is equal to percentage of 100. The measurment can be any where between 0.21 to 1 and this equal to percentage of 21-100%.
Time Frame: 4 hours
Population: The mean of oxygen level (proportion) of all participant after ECALMIST
Measure: Mean (Standard Deviation); unit: Proportion of oxygen saturation
Arm/Group | Surfactant Administration Through Vascular Catheter
Number analyzed (Participants) | 21
Proportion of oxygen saturation | 0.257 (0.084)

13. Secondary Outcome: Needs for Intubation During the Procedure
Description: The needed for interruption or stop of ECALMIST to give PPV (positive pressure ventilation or mechanical ventilation though intubation by ETT (endotracheal intubation)
Time Frame: 10 minutes
Population: The number of preterm infants that needed intubation by ETT (endotracheal intubation) during ECALMIST
Measure: Number; unit: Number of participants
Arm/Group | Surfactant Administration Through Vascular Catheter
Number analyzed (Participants) | 21
Number of participants | 3

ADVERSE EVENTS:
Groups:
- Angiocath Surfactant: Preterm infants from 24 to 34 weeks were received surfactant by using technique called ECALMIST (Early CPAP And Large Volume Minimal Invasive Surfactant)
Arm/Group | Angiocath Surfactant
Serious Adverse Events (participants affected / at risk) | 3/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Angiocath Surfactant (N=21)
Brady cardia (Cardiac disorders) | 1 (21) — Severe brady occurs in 1/21 (14.28%)
de-saturation (Respiratory, thoracic and mediastinal disorders) | 3 (21) — Desaturation bellow 85% for 10 seconds occurs in 3/21 (14.28)

LIMITATIONS AND CAVEATS:
This is non randomized interventional feasibility trial, small sample size and in one center

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No